CLINICAL TRIAL: NCT03311620
Title: TH-112: Pilot Study to Investigate The Diagnostic Yield and Utility of 22g and 19g Endobronchial Ultrasound Transbronchial Needle Aspirate
Brief Title: Pilot Study to Investigate The Diagnostic Yield and Utility of 22g and 19g Endobronchial Ultrasound Transbronchial Needle Aspirate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TH-112
Record Dates: First submitted 2017-10-03; First posted 2017-10-17 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: All abnormal lymph nodes able to be visualized by EBUS will be biopsied with sequential passes until a macroscopic specimen can be seen in the sample container. Each needle size will be used to take consecutive passes until the sample is complete and each pass will consist of 15-20 agitations. The needle size to be used first will be chosen by permuted block randomization scheme by the statistician. After all passes are done with the first needle, the alternate size needle will be used to biopsy the same lymph node. Samples will be placed in separate containers of formalin. Any subsequent lymph nodes in the same patient will be biopsied with the alternate sized needle first. Further, any lung nodules or masses that can be adequately visualized by EBUS where biopsy is clinically indicated will be sampled with both 22g and 19g TBNA needles in the same fashion. However, these lesions will be randomized separately from any lymph nodes biopsied during the case.
Masking Description: The needle size to be used first will be chosen by permuted block randomization scheme by the statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endobronchial ultrasound transbronchial needle aspirate (Other)
  Interventions: Procedure: Endobronchial ultrasound (EBUS) transbronchial needle aspirate (TBNA)

INTERVENTIONS:
Procedure: Endobronchial ultrasound (EBUS) transbronchial needle aspirate (TBNA) — Biopsy samples will be collected from patients scheduled to undergo EBUS TBNA using 19g and 22g needles

SUMMARY:
Needle biopsy samples are routinely collected to evaluate cytomorphology, immunohistochemical markers and for mutational analysis. With regular use of immunotheraputic interventions, needle biospy has become more frequent and requires bigger samples for an increasing battery of tests. There has been no clear consensus on which biopsy needle yields the best biopsy sample. It is unclear if large 19g needle offers better yield than a 22 g needle. Although previous studies comparing 21, 22 and 19g needles have suggested that larger needles yield larger biopsy sizes, conflictng studies have shown that larger biopsies lead to bloodier samples with potentially smaller fragments of tissue, offering no improvement in diagnostic, yield, adequacy or sample size.

This study compares biopsy samples collected using 19g and 22g needles from patients of non small cell lung cancer (NSCLC) scheduled to undergo endobronchial ultrasound (EBUS) and transbroncial needle aspiration (TBNA).

DETAILED DESCRIPTION:
Primary Objective To compare the diagnostic yield of 22g and 19g EBUS transbronchial needle aspirate (TBNA)

Secondary Objectives

1. To compare the sample adequacy of 22g and 19g EBUS TBNA
2. To compare the sample quality of 22g and 19 g EBUS TBNA

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing EBUS TBNA for evaluation of lymphadenopathy, lung nodule or mass
* Patients must have atypical lymph nodes. Atypical lymph nodes are characterized by >10mm in short axis or lymph nodes 5-10mm in short axis with atypical features.
* Age > 18 years.
* Patients must have platelets count > 50,000
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document
* WOCBP must agree not to get pregnant until the day of the procedure

Exclusion Criteria:

* Patients with uncorrectable coagulopathy will be excluded.
* Patients with hemodynamic instability will be excluded
* Patients with refractory hypoxemia will be excluded
* Patients with therapeutic anticoagulant that cannot be held for 2 days before and 1 day after the procedure.
* Patients who are unable to tolerate general anesthesia according to the anesthesiologist
* Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Compare diagnostic yield | 1 year
  Diagnostic yields of 22g and 19g needles will be evaluated by two blinded cytopathologists. Diagnostic yield refers to a specific diagnosis made on the basis of EBUS TBNA samples.

SECONDARY OUTCOMES:
To compare the sample adequacy of 22g and 19g EBUS TBNA | 1 year
  Cytologic/ histologic analysis that determines the amount of sample collected with the two needles by two blinded cytopathologists
To compare the sample quality of 22g and 19 g EBUS TBNA | 1 year
  Sample quality will be examined by two blinded pathologists as to whether the samples contained only tissue or were contaminated with blood

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Manley CJ, Kumar R, Gong Y, Huang M, Wei SS, Nagarathinam R, Haber A, Egleston B, Flieder D, Ehya H. Prospective randomized trial to compare the safety, diagnostic yield and utility of 22-gauge and 19-gauge endobronchial ultrasound transbronchial needle aspirates and processing technique by cytology and histopathology. J Am Soc Cytopathol. 2022 Mar-Apr;11(2):114-121. doi: 10.1016/j.jasc.2021.10.003. Epub 2021 Oct 23. PMID 34896033